CLINICAL TRIAL: NCT07261046
Title: Comparison of the Impact of Two Early Interventions on the Development of Premature Infants: a Clinical Study of Short- and Long-term Effects
Brief Title: Comparison of Two Early Treatments for Premature Babies and Their Effects Over Time
Acronym: PREMOTSENS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Collaborators: Clinique Bouchard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREMOTSENS
Record Dates: First submitted 2025-11-19; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Premature - Weight 1000g-2499g or Gestation of 28-37weeks; Premature Baby 26 to 32 Weeks; Premature Baby 33 to 36 Weeks; Premature Between 32 and 36 Weeks of Amenorrhoea
Keywords: ATVV; multisensory care; preterm outcome; sensory integration; NICU
MeSH Terms: interventions — Touch; Singing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ATVV group (Experimental): The experimental group comprising premature infants receiving ATVV care
  Interventions: Behavioral: ATVV (Auditory, Tactile, Visual and Vestibular stimulation)
- Parental Singing group (Other): The intervention control group comprising premature infants receiving Parental Singing care
  Interventions: Behavioral: Singing
- Control group (No Intervention): The control group comprising full-term infants

INTERVENTIONS:
Behavioral: ATVV (Auditory, Tactile, Visual and Vestibular stimulation) — ATVV consists in providing the infant with multisensory stimulation through massage, talking, eye contact, and gentle rocking.
  Arms: ATVV group
Behavioral: Singing — The singing intervention consists in parents singing softly next to the child's ear.
  Arms: Parental Singing group

SUMMARY:
According to the latest World Health Organization report, prematurity is a major health issue, recognized as a significant vulnerability factor contributing to the emergence of neurodevelopmental disorders. Of the various approaches adopted to limit its consequences, the control of the sensory environment and sensory-focused care are relatively recent. Although a number of sensory care approaches exist, few of them address the different sensory modalities jointly and have been scientifically validated. This research project aims to conduct a study in France on the effectiveness of multisensory ATVV (Auditory, Tactile, Visual, and Vestibular stimulation) treatment using a combination of short- and long-term clinical assessments. The research hypothesis is that ATVV care provided before term age will have a greater impact than "Parental Singing" care on the motor parameters and alertness level of premature infants. Given the importance of motor activity on child development, it is hypothesized here that from term age onwards, the development of children in the ATVV group will be less atypical, or even equivalent to that of the group of full-term infants for most of the parameters evaluated. Furthermore, this normalization of the developmental trajectory will be less pronounced for the "Parental Singing" group. However, the sessions for both treatments (Parental Singing and ATVV) should improve early interactions, sucking, and physiological parameters.

DETAILED DESCRIPTION:
According to a report published by the World Health Organization (WHO) in 2023, 13.4 million infants were born prematurely worldwide in 2020. In France, the 2022 INSERM (Institut national de la santé et de la recherche médicale) report indicates that between 2016 and 2020, the rate of premature births represented 7% of all births and has remained stable for two decades. Prematurity has a significant medical and economic impact in France. It is estimated that the total cost of care (inpatient and outpatient) during the first year of life is approximately €82,000 for infants born before 32 weeks of gestation, compared to an average of only €2,500 for full-term infants. Depending on the degree of prematurity, the outcome for children will vary. Accordingly, the EPIPAGE 2 (Etude épidémiologique sur les petits âges gestationnels) cohort found that 27% of infants born extremely premature, 19% of infants born very premature, and 12% of infants born moderately premature have severe or moderate developmental difficulties (intellectual delay, coordination or neurosensory disorders) during childhood, compared to only 5% of infants born at term. More than a third of premature children also have milder disorders such as neurodevelopmental, behavioral, or sensory disorders. These sensory integration disorders are caused in particular by infections due to the context of premature birth, as well as by the sensory environment of neonatal units, which can lead to central nervous system impairments. Indeed, neonatal units are now known to be "dystimulating" for newborns. Whether due to invasive care, the high-noise environment, antiseptic odors, or high light levels, neonatal units do not provide the same developmental conditions as the intra-uterine environment. As preterm infants do not yet have mature sensory systems, these sensory conditions are greatly disturbing since they cannot be optimally integrated at the cerebral level. These repeated dystimulations induce short-term effects on behavior and physiology, as well as long-term effects such as hypersensitivity, malformations of the sensory cortex, and, more broadly, sensory integration disorders. These cortical alterations manifest as a loss of white matter and a reduced brain size in several brain regions. Several studies have highlighted a link between these sensory integration disorders in premature infants and impaired cognitive development during childhood. Among the approaches implemented in recent years to limit the consequences of prematurity, controlling the sensory environment and providing sensory care for infants are of fundamental importance. To date, there are numerous official recommendations on the subject, such as the document published by the "Care Environment" commission, the report by the "First 1000 Days" commission and that of the "Care Environment" commission, which recommends adapting the hospital environment of neonatal units and taking into account the sensory needs of premature babies. Among the best-known programs for neonatal environmental management is NIDCAP (Newborn Individualized Developmental Care and Assessment Program), which aims to limit sensory dystimulations and adapt care for premature newborns in accordance with their sensory needs. This program recommends that ceiling lights should not exceed a certain brightness threshold and that dimmable ceiling lights should be used. In addition, the noise level of scopes should be reduced whenever possible, care should not be provided while infants are sleeping so as to respect their sleep, and sugar may be administered to limit pain perception. It is also recommended that babies be positioned in their cribs using swaddling blankets, in order to replicate the flexed position that they adopted in their mother's womb. Health authorities also insist on the use of developmental care strategies focused on the sensory abilities of premature infants, making this a key factor in promoting brain plasticity in premature infants. The French National Authority for Health (HAS) also recommends early intervention by psychomotor therapists as a preventive measure on a sensory-perceptual-motor level from the neonatal period onwards. Multisensory care programs have been developed, but only a small proportion are practiced in developmental care in French neonatal units. Sensory-focused treatments mainly center on massage, such as the International Association of Infant Massage program (IAIM), or music therapy. Another commonly used practice is the Kangaroo method, where the parent has skin-to-skin contact with their child. ATVV (Auditory, Tactile, Visual, and Vestibular stimulation) therapy, also known as H-HOPE, is one of the scientifically validated therapies that is not used in France, making it of interest here. In this multisensory treatment, parents are directly involved as they are the ones who implement it, with the support of either pediatric nurses in the US or psychomotor therapists in France. Currently, large-scale training of healthcare professionals is being conducted in the US in order to generalize and systematize this treatment in all neonatal units. This care involves a multisensory stimulation protocol carried out by parents on a daily basis from the moment the premature infant is in stable condition. During 15-minute sessions comprising three codified phases, the parent simultaneously stimulates several of the infant's senses in a coordinated manner, while respecting the infant's rhythm. It is thus possible to distinguish between a phase of oralization/eye contact, a phase of oralization/massage, and a phase of oralization/rocking. The infant's physiological constants and behavioral manifestations are closely monitored. Numerous beneficial effects have been demonstrated, such as a positive effect on infants' alertness, sucking coordination, weight gain, tonic regulation, stress levels, and neurovegetative variables. The treatment also has a positive impact on parents, who are better able to understand the signals emitted by their baby and are more responsive to signs of hunger or sensory dystimulation. However, the link between multisensory care and motor development in premature infants remains understudied. For instance, it is not known when premature infants receive multisensory care, how this affects their motor skills and sensory integration before and after their term age. To date, the mechanisms involved in the link between multisensory integration and movement quality in premature infants remain unexplored. From a methodological point of view, most studies use a control group consisting of full-term infants or premature infants receiving only standard care: the specific effect of "care" is therefore not studied. PREMOTSENS overcomes these methodological limitations by using two comparison groups. The first intervention control group consists of premature infants receiving "Parental Singing" care, where the parent must sing to the infant, and the second control group consists of full-term infants. The choice of a comparison group receiving "Parental Singing" care was made in accordance with the literature. Numerous meta-analyses have shown that singing by parents, with mothers often being the most studied, has benefits for premature infants, including stabilization of certain physiological parameters, more consistent behavior, increased food intake, and analgesic effects during care. Effects on the parent have also been observed, with a decrease in maternal anxiety and improved parent-child synchrony. However, since singing does not require motor skills, no benefits of this treatment have been observed on the motor development of premature infants in either the short or long term, except in a very recent study. This makes the Parental Singing group an ideal comparison group for our experimental group benefiting from the ATVV protocol. Furthermore, most studies have focused on the short-term effects of treatment. In order to provide a more comprehensive analysis, our study will be conducted on two different time scales: a short-term analysis (studying the effects from 34 weeks of gestation to 40 weeks of gestation) and a long-term analysis (studying the effects up to 6 months of corrected age).

ELIGIBILITY:
Inclusion Criteria:

1. For premature infants: birth between 30 and 34 weeks of gestation plus 6 days, and weighing more than 1800 g at the start of the trial.
2. For full-term infants: pregnancy and birth without complications at or after 37 weeks of gestation, with an Apgar score ≥7 at 10 minutes after birth.
3. For parents or legal guardians:

   * Parents over the age of 18
   * Parent agreeing to be filmed with their infant (parent who will be responsible for the treatment)
   * Parents capable of understanding the information document
   * Parent affiliated with or beneficiary of the French social security system
   * Parents who have been informed and have freely given their informed written consent no later than the day of inclusion.

Exclusion Criteria:

1. For premature infants:

   * Birth before 30 weeks of gestation
   * Weight less than 1800 g at the start of the trial
   * Morbidities related to prematurity (necrotizing enterocolitis, cerebral parenchymal damage, stage III and IV intraventricular hemorrhages)
   * Presence of a congenital malformation or chromosomal abnormality
   * Known sensory, motor, or central nervous system impairment
   * Patient receiving non-invasive ventilation at 34 weeks gestational age (CPAP and high-flow nasal cannula)
2. For full-term infants:

   * Birth before 37 weeks gestation
   * Birth with complications
3. For the parent providing the treatment and the infant:

   * Presence of a known sensory, motor, or central nervous system impairment
   * Presence of a congenital condition
   * Presence of psychological distress in the parent
4. For both parents:

   * Under guardianship, conservatorship, or legal protection
   * Situation of extreme psychosocial instability and/or mention of domestic and/or intra-family violence
   * Illicit drug or alcohol use by the mother during the perinatal period
   * Participant is in another study with an ongoing exclusion period during inclusion
   * Involuntary hospitalization

Ages: 0 Weeks to 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Analysis of the long-term impact of ATVV care on premature infants | The primary endpoint will be measured at 6 months corrected age in premature infants, and at 6 months in full-term infants.
  The primary objective is to analyze the long-term impact of ATVV care on premature infants. Motor and cognitive development at 6 months will be compared between premature infants (30 to 34 weeks gestation) receiving ATVV care with premature infants receiving "Singing" care and full-term infants (>37 weeks gestation), using the Bayley Scales of Infant and Toddler Development, 4th Edition (from 16 days to 42 months) and its motor subscore (assessing fine and gross motor skills) and cognition subscore. A subscore (standardized score) ≥ 85 out of 160 in each domain corresponds to typical development.

SECONDARY OUTCOMES:
Motor skills | The outcome is measured between 34 weeks gestational age and 2 months of corrected age.
  Three different motor skills will be measured: spontaneous motor skills, involving general movements and accelerometry (head/forearm/calf); voluntary motor skills, involving Crawliskate in the laboratory with a motion capture system; and oral motor skills, involving sucking a pacifier with a pressure sensor adapted for premature infants.
Overall and communication development | The outcome is measured between 34 weeks gestational age and 2 months of corrected age.
  The outcome is measured using the subscore for the receptive and expressive communication scales, and the ensemble of communication, motor, and cognitive subscores, from the Bayley Scales of Infant and Toddler Development, 4th Edition. A standardized score ≥ 85 out of 160 corresponds to typical development.
Multisensory integration | The outcome is measured between 34 weeks gestational age and 2 months of corrected age.
  A visuo-vestibular conflict paradigm using a device that measures head acceleration of the infant.
Level of alertness | The outcome is measured between 34 weeks gestational age and 2 months of corrected age.
  Alertness is evaluated on the Prechtl assessment scale, comprising 5 levels: quiet sleep; active/restless sleep; quiet wakefulness; restless wakefulness; and agitation.
Precocious interactions | The outcome is measured between 34 weeks gestational age and 2 months of corrected age.
  The outcome is measured using a scale of mutual dyadic (parent-child) interactions from the Dyadic Mutuality Code (Censuello) that ranks 6 items as present or absent: mutual attention; positive affects; interactional turn-taking; maternal pauses; clarity of infant cues; and maternal sensitivity and responsiveness.
Parenting stress | The outcome is measured at 2 months of corrected age.
  The outcome is evaluated according to the PSI-4-SF parenting stress index questionnaire, which divides 36 items into the following subscales: parenting stress; dysfunctional parent-child interaction; and difficult child. Each item is rated from 1 (strongly disagree) to 5 (strongly agree), to determine whether parental stress is low, fair or elevated.
Heart rate | The outcome measure will be provided by the parent from 34 weeks gestational age to term equivalent age.
  Infants in the prenatal service are monitored for heart rate. Heart rate values will be read by parents from the monitor screen, once per minute for five minutes. The expected value for premature infants is between 130-170 beats per minutes.
Respiratory rate | The outcome measure will be provided by the parent from 34 weeks gestational age to term equivalent age.
  Infants in the prenatal service are monitored for respiratory rate. Respiratory rate will be read by parents from the monitor screen, once per minute for five minutes. The expected value for premature infants is approximately 50 cycles/minute.
Oxygen saturation | The outcome measure will be provided by the parent from 34 weeks gestational age to term equivalent age.
  Infants in the prenatal service are monitored for oxygen saturation. Oxygen saturation will be read by parents from the monitor screen, once per minute for five minutes. The expected value for premature infants is between 85-95%.
Weight | Weight will be recorded at 2 and 6 months corrected age.
  Weight will be taken from medical records. Weight gain (kg) will be monitored for each infant.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinique Bouchard, Marseille
  - Hopital Saint-Joseph, Marseille